CLINICAL TRIAL: NCT05342831
Title: The Effect of Biological Nutrition Technique Which is Used in Initiation of Breastfeeding in Primiparas on Breastfeeding Success and on Self-Efficacy: A Randomized Controlled Study
Brief Title: Biological Nutrition Technique Which is Used in Initiation of Breastfeeding
Acronym: BNTPBSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hatice Gul OZTAS (Other)
Responsible Party: Sponsor-Investigator, Hatice Gul OZTAS, Asst. Prof. Dr., Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KSUHATİCEGULOZTAS001
Record Dates: First submitted 2022-04-04; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Breast Feeding; Self Efficacy
Keywords: Primiparous; Midwifery
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: experimental group (Experimental): Biological Nutrition Technique
  Interventions: Other: Biological Nutrition Technique
- Assigned Interventions (No Intervention): standard care group

INTERVENTIONS:
Other: Biological Nutrition Technique — Biological nutrition technique woman trying Biological feeding technique was applied after each breastfeeding. Breastfeeding self-efficacy and breastfeeding success were assessed at regular intervals.
  Arms: Experimental: experimental group

SUMMARY:
Aim: This research was conducted with the purpose of determining the effect of biological nurturing technique used for starting breastfeeding in primipara on breastfeeding success and self-efficacy.

Material and Method: This randomized controlled study was conducted with 130 mothers who had a cesarean section in a public hospital located in Southeast Turkey (65 experimental, 65 control).

DETAILED DESCRIPTION:
Aim: This research was conducted with the purpose of determining the effect of biological nurturing technique used for starting breastfeeding in primipara on breastfeeding success and self-efficacy.

Material and Method: This randomized controlled study was conducted with 130 mothers who had a cesarean section in a public hospital located in Southeast Turkey (65 experimental, 65 control). The mothers in the control group received routine hospital care. The mothers in the experimental group were taught the biological nurturing technique after the first breastfeeding and breastfeeding was provided according to the technique during the hospitalization. Pre-test data were obtained by applying LATCH and BSES-SF to the mothers in the experimental and control groups at the 1st hour after the first breastfeeding. LATCH was re-administered at the end of the 8th and 24th hour postpartum. Post-test data were obtained by administering LATCH and BSES at the end of the 48th hour postpartum.In statistical analysis; count, percentage distribution, arithmetic average, chi-square test, standard deviation, t-test in dependent and independent groups and ANOVA analysis in repeated measurements were used.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years and older,
* Having a full-term, single and healthy newborn,
* Having no known health problems
* Having no general anesthesia
* Implementation of planned cesarean delivery,
* Primiparous women who do not have a condition that prevents breastfeeding. Inclusion criteria of the research for infants

Exclusion Criteria:

• Women with a risky pregnancy diagnosis (such as preeclampsia, placenta previa, gestational diabetes)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
First Measurement:LATCH | Measurement at the second encounter (first 24 hours after birth) for each group.
  Observation and evaluation of mothers' breastfeeding success is measured using the LATCH scale.The LATCH Breastfeeding Diagnostic and Evaluation Scale is a scale filled by the researcher through observation.
  L: (Latch on the brest)) A: (Audible Swallowing) T: (Type of Nipple) C: (Comfort of Breast/ Nipple) H: (Hold/ Position)
  LATCH consists of the combination of the first letters of the English equivalent of the five criteria defined above. Each item is evaluated between 0-2 points. The lowest score that can be obtained from the entire scale is 0 and the highest score is 10. The scale has no breakpoints. The low score on the scale indicates the need for active intervention, support and follow-up after discharge in breastfeeding. The higher the LATCH Breastfeeding Diagnosis and Evaluation Scale score, the higher the success of breastfeeding.
Second Measurement:Breastfeeding Self-Efficacy Scale Çeviri sonuçları Breastfeeding Self-Efficacy Scale | Measurement for each group at the third encounter (2th day after birth).
  Breastfeeding self-efficacy levels and breastfeeding self-confidence of mothers are measured with the breastfeeding self-efficacy scale. The Breastfeeding Self-Efficacy Scale (short form) consists of 14 items that measure the mother's breastfeeding self-efficacy. The maximum score that can be obtained from the scale is 70, and the minimum score is 14. High scores from the scale indicate high breastfeeding self-efficacy. The scale is 5-point Likert type; 1 = Not at all sure, 2 = Not so sure, 3 = Sometimes I'm sure, 4 = I'm sure, 5 = I'm very sure.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Gül Öztaş, Principal Investigator — KahramanmaraşISU; Yeşim Aksoy Derya, Study Director — İnönü University
Locations (1):
- Kahramanmaraş ISU, Kahramanmaraş, K.Maraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
we don't share individual participant data with other researchers

REFERENCES:
- [Result] Milinco M, Travan L, Cattaneo A, Knowles A, Sola MV, Causin E, Cortivo C, Degrassi M, Di Tommaso F, Verardi G, Dipietro L, Piazza M, Scolz S, Rossetto M, Ronfani L; Trieste BN (Biological Nurturing) Investigators. Effectiveness of biological nurturing on early breastfeeding problems: a randomized controlled trial. Int Breastfeed J. 2020 Apr 5;15(1):21. doi: 10.1186/s13006-020-00261-4. PMID 32248838
- See also: Effectiveness of biological nurturing on early breastfeeding problems: a randomized controlled trial — https://scholar.google.com/scholar?hl=tr&as_sdt=0%2C5&q=Effectiveness+of+biological+nurturing+on+early+breastfeeding+problems%3A+a+randomized+controlled+trial&btnG